CLINICAL TRIAL: NCT06696066
Title: Pilot Evaluation of a Peer Recovery Support Program Adapted to Target Retention in Clinic-based Medication for Opioid Use Disorder Treatment
Brief Title: PEERS Pilot: Peer Recovery Support Program to Support Engagement in Medication for Opioid Use Disorder
Acronym: PEERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); UConn Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0862; 1R61DA059880 (NIH)
Record Dates: First submitted 2024-11-18; First posted 2024-11-19 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Opioid Use Disorder
Keywords: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer Recovery Support Pilot Program Implementation and Assessment (Experimental): Participants will be offered services from a certified recovery specialist (i.e., the Peer Recovery Support program). This will entail a CRS meeting one-on-one with the patient at regular intervals (e.g., weekly) to provide support to the participant for a 6-month period. CRS services are patient-centered and driven by a patient's own recovery goals, thus the frequency, timing, duration, modality (in-person, phone), and location of meetings (in the clinic or in a community setting such as a coffeeshop) are flexible and determined collaboratively by the CRS and patient.
  Interventions: Behavioral: PRS Program

INTERVENTIONS:
Behavioral: PRS Program — The Peer Recovery Support program will be delivered by a certified recovery specialist (CRS) over the course of 6-months. The CRS will provide supportive care to the participant during their initial 6-months of MOUD treatment to increase patient engagement in their treatment. The CRS may provide emotional support; help participants to identify their recovery assets, goals, and barriers; guide participants in creating a recovery plan; help participants to increase their coping skills; and assist participants in connecting to community and recovery resources.

SUMMARY:
The goal of this pilot study is to evaluate the feasibility and acceptability of implementing a peer recovery support program to support patient engagement in medication treatment for opioid use disorder (MOUD). The program, entitled "Promoting Enhanced Engagement through Recovery Support" (PEERS) was developed in collaboration with community and clinical partners for the MOUD outpatient setting. Information gathered during this pilot study will inform refinements to the program and study components for a future clinical trial that will evaluate the effectiveness of the peer recovery support program in increasing patient retention in MOUD.

The investigators will recruit 12 participants to the pilot study, all of whom will receive the PEERS program. The study will take place in Geisinger outpatient addiction treatment clinics in northeast Pennsylvania. Patients initiating MOUD treatment at one of the clinics will be eligible for participation, and will be recruited via email, patient portal messages, and phone. Each participant will receive the PEERS program, entailing regular sessions with a Certified Recovery Specialist (CRS) for 6 months. Participants will also be asked to complete assessments at baseline and 12 weeks and will be invited to provide qualitative feedback on their experience with the program through an interview conducted between 8-12 weeks. As the focus of the pilot pertains to the feasibility and acceptability of the program and the study components, study outcomes focus on participant engagement in and acceptance of the program, CRS fidelity to the program, barriers to implementation, and feasibility of data collection.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years of age
* Initiated medication for opioid use disorder at a Geisinger outpatient addiction treatment clinic within the past 45 days
* Willing to participate in the Peer Recovery Support program
* Able and willing to provide consent

Exclusion Criteria:

* Received medication for opioid use disorder at a Geisinger outpatient addiction treatment clinic in the 90 days prior to the treatment initiation date
* Not proficient in English

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Feasibility - participant engagement in the peer recovery support program | Baseline to 12 weeks
  Average number of sessions participants attended with the Certified Recovery Specialist
Acceptability - participant acceptability of the peer recovery support program | 8 to 12 weeks
  Qualitative responses from participant interviews regarding the helpfulness of the program in their recovery from opioid use disorder
Acceptability - participant alliance with Certified Recovery Specialist | 12 weeks
  Participants' average scores for the Scales for Participant Alliance with Recovery Coach (SPARC-2)
Fidelity - Certified Recovery Specialist fidelity to peer recovery support program components | Baseline to 6 months
  Appropriate delivery of program components during participant sessions, as measured with a fidelity checklist
Feasibility - barriers faced by Certified Recovery Specialist in delivering peer recovery support program | Baseline to 6 months
  Log of qualitative feedback from Certified Recovery Specialist regarding the barriers to program delivery
Feasibility - peer recovery support program integration into clinical setting | 6 months
  A short survey will assess clinic staff's perceptions of the integration of the Certified Recovery Specialist into the clinic flow

SECONDARY OUTCOMES:
Feasibility - feasibility of assessment completion | Baseline, 12 weeks
  Completion proportion of baseline and follow-up assessments by participants. Average participant rating of comprehensibility and acceptability of length of assessments
Acceptability - acceptability of incentives | Baseline, 12 weeks
  Average participant rating of the acceptability of incentive amounts and gift card types received for assessment completion

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Poulsen, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health, Danville, Pennsylvania, United States

DOCUMENTS (1):
  • Informed Consent Form (2025-02-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT06696066/ICF_000.pdf